CLINICAL TRIAL: NCT04684212
Title: Can the Lambre Device Occlude IRRegular And Large Appendages in Patients With Non-Valvular AF: The CORRAL-AF Study
Brief Title: Can the Lambre Device Occlude IRRegular And Large Appendages in Patients With Non-Valvular AF
Acronym: CORRAL-AF
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Lack of Funding
Sponsor: Brian O'Neill MD (Other)
Collaborators: Lifetech Scientific (Shenzhen) Co., Ltd. (Industry)
Responsible Party: Sponsor-Investigator, Brian O'Neill MD, Director of Interventional Cardiology Research, Henry Ford Health System
Organization: Henry Ford Health System (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: G-200316
Record Dates: First submitted 2020-12-17; First posted 2020-12-24 (Actual); Last update posted 2025-11-04 (Actual); Status verified 2025-10

CONDITIONS: Atrial Fibrillation; Left Atrial Appendage Thrombosis; CVA
Keywords: LAMBRE device; Left Atrial Appendage Occlusion device; CVA prevention; Atrial Fibrillation; Cardiovascular angiography; Anti-coagulation management; Thromboembolism; nonvalvular atrial fibrillation; non-pharmacological alternative; Thrombosis
MeSH Terms: conditions — Atrial Fibrillation; Thromboembolism; Thrombosis | interventions — Warfarin; Dabigatran; Rivaroxaban; apixaban; edoxaban; betrixaban

STUDY DESIGN:
Intervention Model Description: This prospective, randomized, multicenter study will enroll 2,931 subjects (2706 randomized subjects, 225 roll-in subjects) at up to 75 investigational sites in the United States.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (3):
- Device Arm (Experimental): The LAmbre PlusTM Left Atrial Appendage Closure System (LAmbre device)
  Interventions: Device: LAmbre PlusTM Left Atrial Appendage Closure System
- Control Arm (Active Comparator): Market approved oral anticoagulation (OAC)
  Interventions: Drug: Market approved oral anticoagulation (OAC), such as warfarin (Coumadin), dabigatran (Pradaxa), rivaroxaban (Xarelto), apixiban (Eliquis), edoxaban (Savaysa), or betrixaban (Bevyxxa)
- Roll-in Arm (Other): 225 roll-in subjects
  Interventions: Device: LAmbre PlusTM Left Atrial Appendage Closure System

INTERVENTIONS:
Device: LAmbre PlusTM Left Atrial Appendage Closure System — The LAmbre Plus device is a self-expanding occluder, composed of a distal Umbrella and a proximal Cover laser welded together, delivered percutaneously via femoral venous access and trans-septal puncture. The distal Umbrella consists of an elastic nitinol frame and outer PET membrane, and has circumferential anchors to secure the occluder to the left atrial appendage (LAA) wall. The proximal Cover is a disc of elastic nitinol mesh, which seals the orifice of the LAA and minimizes thrombus formation, and includes a PET membrane to prevent the passage of blood into the LAA after implantation.
  Other Names: LAmbre device
  Arms: Device Arm; Roll-in Arm
Drug: Market approved oral anticoagulation (OAC), such as warfarin (Coumadin), dabigatran (Pradaxa), rivaroxaban (Xarelto), apixiban (Eliquis), edoxaban (Savaysa), or betrixaban (Bevyxxa) — Continuation of market approved OAC drug.
  Other Names: OAC
  Arms: Control Arm

SUMMARY:
The primary objective is to demonstrate the safety and efficacy of the implantation of the LAmbre PlusTM device in patients with large or irregularly shaped appendages with non-valvular atrial fibrillation who are at increased risk for stroke and systemic embolism compared to oral anticoagulation (OAC).

DETAILED DESCRIPTION:
This prospective, randomized, multicenter study will enroll 2,931 subjects (2706 randomized subjects, 225 roll-in subjects) at up to 75 investigational sites in the United States. Patients presenting with non-valvular atrial fibrillation who are at increased risk for stroke and systemic embolism based on CHA2DS2-VASc scores, and who are recommended for oral anticoagulation therapy but have an appropriate rationale to seek a non-pharmacologic alternative to oral anticoagulation, and who meet all eligibility criteria will be enrolled in the study.

Subjects will have clinical follow-up in-hospital and at 45 days, 6 months, 12 months, and annually up to 5-years. CT/Imaging or Transesophageal echocardiographic (TEE) follow-up will occur at 45 days and TEE at 1-year.

The LAmbre PlusTM Left Atrial Appendage (LAA) Closure System is intended to reduce the risk of thromboembolism from the left atrial appendage (LAA) in patients with nonvalvular atrial fibrillation who:

* Are at increased risk for stroke and systemic embolism based on CHADS2 or CHA2DS2-VASc scores and are recommended for oral anticoagulation (OAC) therapy; AND
* Are deemed by their physician to be suitable for OAC; AND
* Have an appropriate rationale to seek a non-pharmacological alternative to OAC, taking into account the safety and effectiveness of the device compared to OAC

ELIGIBILITY:
Potential subjects must meet ALL of the following criteria to be eligible for inclusion in the study:

Inclusion Criteria:

1. The patient is a male or non-pregnant female ≥18 years of age
2. The patient has documented paroxysmal, persistent, or permanent non-valvular atrial fibrillation or flutter
3. The patient has a CHADS2 score ≥ 2 or a CHA2DS2-VASc score of ≥ 3, and is recommended for oral anticoagulation therapy
4. The patient is deemed by their physician to be suitable for short-term OAC, but there is an appropriate rationale for seeking a non-pharmacologic alternative to oral anticoagulation
5. The patient is deemed suitable for LAA closure in a shared decision model with a non-implanting physician
6. The patient is willing and able to comply with protocol-specified treatment and follow-up evaluations
7. The patient (or his or her legally authorized representative) has been informed of the nature of the study, agrees to its provisions, and has been provided written informed consent approved by the appropriate Institutional Review Board (IRB) or Ethics Committee (EC)

Potential subjects will be excluded if ANY of the following conditions apply:

Exclusion Criteria:

1. Pregnant or nursing patients and those who plan pregnancy in the period up to 1 year following index procedure. Female patients of childbearing potential must have a negative pregnancy test done within 7 days prior to index procedure per site standard test
2. Patients with atrial fibrillation that is defined by a single occurrence, or that is transient or reversible (e.g., secondary to CABG, an interventional procedure, pneumonia, or hyperthyroidism)
3. Patients who require long-term anticoagulation/DAPT for a condition other than atrial fibrillation
4. Patients not suitable for short term oral anti-coagulation (including due to bleeding diathesis or coagulopathy or absolute contraindication to OAC or DAPT ) or who will refuse transfusion
5. Patients with rheumatic mitral valve disease, known severe aortic stenosis requiring surgical or percutaneous valve replacement, or existing mechanical valve prosthesis
6. Active infection with bacteremia
7. Known hypersensitivity or contraindication to aspirin, clopidogrel, heparin/bivalirudin, any device material or component (nitinol, nickel, titanium, PET), and/or contrast sensitivity that cannot be adequately pre-medicated
8. Anatomic conditions that would prevent performance of the LAA occlusion procedure (e.g., prior atrial septal defect [ASD] or patient foramen ovale [PFO] surgical repair or implanted closure device, or obliterated left atrial appendage)
9. Recent (within 30 days pre-procedure) or planned (within 60 days post procedure) cardiac or non-cardiac interventional or surgical procedure (e.g., cardioversion, ablation, percutaneous coronary intervention, cataract surgery, etc.)
10. Recent (within 90 days pre-procedure) stroke, transient ischemic attack, or myocardial infarction
11. Severe heart failure (New York Heart Association Class IV)
12. Known asymptomatic carotid artery disease with>70% diameter stenosis OR symptomatic carotid disease (>50% diameter stenosis with ipsilateral stroke or TIA). Subjects with prior carotid endarterectomy or carotid stent placement may be enrolled, provided that known diameter stenosis is <50%.
13. Past or pending heart or any other organ transplant, or on the waiting list for any organ transplant
14. Current participation in another investigational drug or device study
15. Size of the left atrial appendage at the LAmbre Plus defined landing zone within outside the manufactures recommendations (Table 2.)
16. Patients with an indication for chronic P2Y12 platelet inhibition therapy
17. Patients who are unable to undergo CT scan

Echocardiographic Exclusion Criteria

1. Left atrial appendage anatomy may accommodate implantation of the WATCHMAN device, according to IFU by size.
2. LVEF <25%
3. Intracardiac thrombus or dense spontaneous echo contrast, as visualized by TEE within 2 days prior to implant
4. Presence of a high-risk patent foramen ovale (PFO), defined as an atrial septal aneurysm (excursion >15 mm or length >15 mm) or large shunt (early, within 3 beats and/or substantial passage of bubbles)
5. Moderate or severe mitral valve stenosis (mitral valve area <1.5 cm2)
6. Complex atheroma with mobile plaque of the descending aorta and/or aortic arch (Grade 4 or higher)
7. Presence of an intracardiac tumor

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2024-06-01 (Estimated); Primary Completion 2024-06-01 (Estimated); Study Completion 2024-07-11 (Actual)

PRIMARY OUTCOMES:
Composite of time to first occurrence of stroke, cardiovascular death, or clinically relevant major or non-major bleeding events | through study completion, up to 5 years
  Defined as composite of: First occurrence of stroke defined by NeuroARC; Cardiovascular death defined as any death due to proximate cause (e.g., MI, low-output failure, fatal arrhythmia), unwitnessed death and death of unknown cause, and all procedure related deaths, including those related to concomitant treatment; Clinically relevant major or non-major bleeding events defined by hemoglobin of ≥2.0 g/dl during a 24-h period, transfusion of ≥2 units of packed red cells, bleeding at a critical site (intracranial, intraspinal, intraocular, pericardial, intramuscular with compartment syndrome, or retroperitoneal), or fatal bleeding
Composite of time to first occurrence of ischemic stroke or systemic embolism | through study completion, up to of 5 years
  Defined as composite of: First occurrence of ischemic stroke defined by NeuroARC; Systemic embolization defined as acute vascular insufficiency or occlusion of the extremities or any non-CNS organ associated with clinical, imaging, surgical/autopsy evidence of arterial occlusion in the absence of other likely mechanism (e.g. trauma, atherosclerosis, or instrumentation). When there is presence of prior peripheral artery disease, angiographic or surgical or autopsy evidence is required to show abrupt arterial occlusion.
Overall safety | 12 months
  Overall safety is defined as the composite of: Major procedure-related complications, defined as the composite of cardiac perforation, pericardial effusion with tamponade, device embolization, and major vascular complications (adjudicated by the independent Clinical Events Committee as related to the study device or procedure); AND Major adverse events, defined as all death, all stroke and major bleeding as compared to OAC

SECONDARY OUTCOMES:
Mortality | 45 days, 6 months, 12 months, 5 years
  Death classified as cardiovascular or non-cardiovascular and reported cumulatively and individually
Myocardial Infarction | 45 days, 6 months, 12 months, 5 years
  Occurrence of MI defined by modified Third Universal Definition, which will be adjudicated and classified by an independent Clinical Events Committee (CEC)
Peri-Procedural Stroke | 30 days
  Occurrence of peri-procedural stroke defined as Overt CNS Injury (NeuroARC defined)
Bleeding Complications | 45 days, 6 months, 12 months, 5 years
  Occurrence of bleeding complications evaluated as major bleeding (BARC Type ≥3); major and minor bleeding (BARC ≥2) and its components by BARC Type
Major Procedure-Related Complications | 45 days
  Occurrence of major procedure-related complications, defined as the composite of cardiac perforation, pericardial effusion with tamponade, ischemic stroke (NeuroARC defined), device embolization, major vascular complications (VARC 3 defined), and major bleeding
Vascular Complications | 45 days, 6 months, 12 months, 5 years
  Occurrence of Vascular complications (VARC 3 defined)
Embolic events | 45 days, 6 months, 12 months, 5 years
  Occurrence of embolic events, defined as the composite of ischemic stroke (NeuroARC defined) and systemic embolization
Ischemic Stroke | 45 days, 6 months, 12 months, 5 years
  Occurrence of ischemic stroke (NeuroARC defined)
Systemic embolization | 45 days, 6 months, 12 months, 5 years
  Occurrence of systemic embolization defined by acute vascular insufficiency or occlusion of the extremities or any non-CNS organ associated with clinical, imaging, surgical/autopsy evidence of arterial occlusion in the absence of other likely mechanism (e.g. trauma, atherosclerosis, or instrumentation). When there is presence of prior peripheral artery disease, angiographic or surgical or autopsy evidence is required to show abrupt arterial occlusion.
All CNS injury and dysfunction | 45 days, 6 months, 12 months, 5 years
  Occurrence of all CNS injury and dysfunction (NeuroARC defined)
Technical success | within 24 hours Post-procedure
  Technical success is defined as successful implantation (acceptable device position, stability, and LAA seal) with the assigned device
Closure success | 45 days
  Closure success is defined as technical success followed by successful LAA closure (complete LAA closure or peri-device residual jet <5 mm in width by TEE/Imaging or CT)
Procedural Success | 7 days Post-procedure
  Procedural success is defined as technical success without major procedure-related complications
Total Procedural Time | within 24 hours Post-procedure
  Total procedural time is defined as time elapsed between first venous access and removal of the last catheter from the venous access sheath
Device Thrombosis | 45 days, 6 months, 12 months, 5 years
  Occurrence of device thrombosis

CONTACTS AND LOCATIONS:
Overall Officials: Brian O'Neill, MD, Principal Investigator — Henry Ford Health System
Locations (1):
- Henry Ford Hospital, Detroit, Michigan, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Mandalenakis Z, Von Koch L, Eriksson H, Dellborg M, Caidahl K, Welin L, Rosengren A, Hansson PO. The risk of atrial fibrillation in the general male population: a lifetime follow-up of 50-year-old men. Europace. 2015 Jul;17(7):1018-22. doi: 10.1093/europace/euv036. Epub 2015 Apr 4. PMID 25842274
- [Background] Heeringa J, van der Kuip DA, Hofman A, Kors JA, van Herpen G, Stricker BH, Stijnen T, Lip GY, Witteman JC. Prevalence, incidence and lifetime risk of atrial fibrillation: the Rotterdam study. Eur Heart J. 2006 Apr;27(8):949-53. doi: 10.1093/eurheartj/ehi825. Epub 2006 Mar 9. PMID 16527828
- [Background] Go AS, Hylek EM, Phillips KA, Chang Y, Henault LE, Selby JV, Singer DE. Prevalence of diagnosed atrial fibrillation in adults: national implications for rhythm management and stroke prevention: the AnTicoagulation and Risk Factors in Atrial Fibrillation (ATRIA) Study. JAMA. 2001 May 9;285(18):2370-5. doi: 10.1001/jama.285.18.2370. PMID 11343485
- [Background] Dewland TA, Olgin JE, Vittinghoff E, Marcus GM. Incident atrial fibrillation among Asians, Hispanics, blacks, and whites. Circulation. 2013 Dec 3;128(23):2470-7. doi: 10.1161/CIRCULATIONAHA.113.002449. Epub 2013 Oct 8. PMID 24103419
- [Background] Lau DH, Nattel S, Kalman JM, Sanders P. Modifiable Risk Factors and Atrial Fibrillation. Circulation. 2017 Aug 8;136(6):583-596. doi: 10.1161/CIRCULATIONAHA.116.023163. PMID 28784826
- [Background] Wolf PA, Abbott RD, Kannel WB. Atrial fibrillation as an independent risk factor for stroke: the Framingham Study. Stroke. 1991 Aug;22(8):983-8. doi: 10.1161/01.str.22.8.983. PMID 1866765
- [Background] Stewart S, Hart CL, Hole DJ, McMurray JJ. A population-based study of the long-term risks associated with atrial fibrillation: 20-year follow-up of the Renfrew/Paisley study. Am J Med. 2002 Oct 1;113(5):359-64. doi: 10.1016/s0002-9343(02)01236-6. PMID 12401529
- [Background] Kong B, Liu Y, Huang H, Jiang H, Huang C. Left atrial appendage closure for thromboembolism prevention in patients with atrial fibrillation: advances and perspectives. J Thorac Dis. 2015 Feb;7(2):199-203. doi: 10.3978/j.issn.2072-1439.2015.01.20. PMID 25713737
- [Background] Hart RG, Pearce LA, Aguilar MI. Meta-analysis: antithrombotic therapy to prevent stroke in patients who have nonvalvular atrial fibrillation. Ann Intern Med. 2007 Jun 19;146(12):857-67. doi: 10.7326/0003-4819-146-12-200706190-00007. PMID 17577005
- [Background] January CT, Wann LS, Alpert JS, Calkins H, Cigarroa JE, Cleveland JC Jr, Conti JB, Ellinor PT, Ezekowitz MD, Field ME, Murray KT, Sacco RL, Stevenson WG, Tchou PJ, Tracy CM, Yancy CW; American College of Cardiology/American Heart Association Task Force on Practice Guidelines. 2014 AHA/ACC/HRS guideline for the management of patients with atrial fibrillation: a report of the American College of Cardiology/American Heart Association Task Force on Practice Guidelines and the Heart Rhythm Society. J Am Coll Cardiol. 2014 Dec 2;64(21):e1-76. doi: 10.1016/j.jacc.2014.03.022. Epub 2014 Mar 28. No abstract available. PMID 24685669
- [Background] Gage BF, van Walraven C, Pearce L, Hart RG, Koudstaal PJ, Boode BS, Petersen P. Selecting patients with atrial fibrillation for anticoagulation: stroke risk stratification in patients taking aspirin. Circulation. 2004 Oct 19;110(16):2287-92. doi: 10.1161/01.CIR.0000145172.55640.93. Epub 2004 Oct 11. PMID 15477396
- [Background] Lip GY, Nieuwlaat R, Pisters R, Lane DA, Crijns HJ. Refining clinical risk stratification for predicting stroke and thromboembolism in atrial fibrillation using a novel risk factor-based approach: the euro heart survey on atrial fibrillation. Chest. 2010 Feb;137(2):263-72. doi: 10.1378/chest.09-1584. Epub 2009 Sep 17. PMID 19762550
- [Background] Pisters R, Lane DA, Nieuwlaat R, de Vos CB, Crijns HJ, Lip GY. A novel user-friendly score (HAS-BLED) to assess 1-year risk of major bleeding in patients with atrial fibrillation: the Euro Heart Survey. Chest. 2010 Nov;138(5):1093-100. doi: 10.1378/chest.10-0134. Epub 2010 Mar 18. PMID 20299623
- [Background] Brass LM, Krumholz HM, Scinto JM, Radford M. Warfarin use among patients with atrial fibrillation. Stroke. 1997 Dec;28(12):2382-9. doi: 10.1161/01.str.28.12.2382. PMID 9412618
- [Background] Chan PS, Maddox TM, Tang F, Spinler S, Spertus JA. Practice-level variation in warfarin use among outpatients with atrial fibrillation (from the NCDR PINNACLE program). Am J Cardiol. 2011 Oct 15;108(8):1136-40. doi: 10.1016/j.amjcard.2011.06.017. Epub 2011 Jul 26. PMID 21798501
- [Background] Go AS, Hylek EM, Borowsky LH, Phillips KA, Selby JV, Singer DE. Warfarin use among ambulatory patients with nonvalvular atrial fibrillation: the anticoagulation and risk factors in atrial fibrillation (ATRIA) study. Ann Intern Med. 1999 Dec 21;131(12):927-34. doi: 10.7326/0003-4819-131-12-199912210-00004. PMID 10610643
- [Background] Birman-Deych E, Radford MJ, Nilasena DS, Gage BF. Use and effectiveness of warfarin in Medicare beneficiaries with atrial fibrillation. Stroke. 2006 Apr;37(4):1070-4. doi: 10.1161/01.STR.0000208294.46968.a4. Epub 2006 Mar 9. PMID 16528001
- [Background] Mant J, Hobbs FD, Fletcher K, Roalfe A, Fitzmaurice D, Lip GY, Murray E; BAFTA investigators; Midland Research Practices Network (MidReC). Warfarin versus aspirin for stroke prevention in an elderly community population with atrial fibrillation (the Birmingham Atrial Fibrillation Treatment of the Aged Study, BAFTA): a randomised controlled trial. Lancet. 2007 Aug 11;370(9586):493-503. doi: 10.1016/S0140-6736(07)61233-1. PMID 17693178
- [Background] Broderick JP, Bonomo JB, Kissela BM, Khoury JC, Moomaw CJ, Alwell K, Woo D, Flaherty ML, Khatri P, Adeoye O, Ferioli S, Kleindorfer DO. Withdrawal of antithrombotic agents and its impact on ischemic stroke occurrence. Stroke. 2011 Sep;42(9):2509-14. doi: 10.1161/STROKEAHA.110.611905. Epub 2011 Jun 30. PMID 21719769
- [Background] Patel MR, Mahaffey KW, Garg J, Pan G, Singer DE, Hacke W, Breithardt G, Halperin JL, Hankey GJ, Piccini JP, Becker RC, Nessel CC, Paolini JF, Berkowitz SD, Fox KA, Califf RM; ROCKET AF Investigators. Rivaroxaban versus warfarin in nonvalvular atrial fibrillation. N Engl J Med. 2011 Sep 8;365(10):883-91. doi: 10.1056/NEJMoa1009638. Epub 2011 Aug 10. PMID 21830957
- [Background] Connolly SJ, Ezekowitz MD, Yusuf S, Eikelboom J, Oldgren J, Parekh A, Pogue J, Reilly PA, Themeles E, Varrone J, Wang S, Alings M, Xavier D, Zhu J, Diaz R, Lewis BS, Darius H, Diener HC, Joyner CD, Wallentin L; RE-LY Steering Committee and Investigators. Dabigatran versus warfarin in patients with atrial fibrillation. N Engl J Med. 2009 Sep 17;361(12):1139-51. doi: 10.1056/NEJMoa0905561. Epub 2009 Aug 30. PMID 19717844
- [Background] Granger CB, Alexander JH, McMurray JJ, Lopes RD, Hylek EM, Hanna M, Al-Khalidi HR, Ansell J, Atar D, Avezum A, Bahit MC, Diaz R, Easton JD, Ezekowitz JA, Flaker G, Garcia D, Geraldes M, Gersh BJ, Golitsyn S, Goto S, Hermosillo AG, Hohnloser SH, Horowitz J, Mohan P, Jansky P, Lewis BS, Lopez-Sendon JL, Pais P, Parkhomenko A, Verheugt FW, Zhu J, Wallentin L; ARISTOTLE Committees and Investigators. Apixaban versus warfarin in patients with atrial fibrillation. N Engl J Med. 2011 Sep 15;365(11):981-92. doi: 10.1056/NEJMoa1107039. Epub 2011 Aug 27. PMID 21870978
- [Background] Kalra L, Yu G, Perez I, Lakhani A, Donaldson N. Prospective cohort study to determine if trial efficacy of anticoagulation for stroke prevention in atrial fibrillation translates into clinical effectiveness. BMJ. 2000 May 6;320(7244):1236-9. doi: 10.1136/bmj.320.7244.1236. PMID 10797031
- [Background] Ono A, Fujita T. Low-intensity anticoagulation for stroke prevention in elderly patients with atrial fibrillation: efficacy and safety in actual clinical practice. J Clin Neurosci. 2005 Nov;12(8):891-4. doi: 10.1016/j.jocn.2004.10.011. Epub 2005 Nov 3. PMID 16271478
- [Background] Ruiz Ortiz M, Romo Penas E, Franco Zapata MF, Mesa Rubio D, Anguita Sanchez M, Lopez Granados A, Arizon del Prado JM, Valles Belsue F. Oral anticoagulation in patients aged 75 years or older with chronic non-valvar atrial fibrillation: effectiveness and safety in daily clinical practice. Heart. 2005 Sep;91(9):1225-6. doi: 10.1136/hrt.2004.050831. No abstract available. PMID 16103572
- [Background] Katz ES, Tsiamtsiouris T, Applebaum RM, Schwartzbard A, Tunick PA, Kronzon I. Surgical left atrial appendage ligation is frequently incomplete: a transesophageal echocardiograhic study. J Am Coll Cardiol. 2000 Aug;36(2):468-71. doi: 10.1016/s0735-1097(00)00765-8. PMID 10933359
- [Background] Holmes DR, Reddy VY, Turi ZG, Doshi SK, Sievert H, Buchbinder M, Mullin CM, Sick P; PROTECT AF Investigators. Percutaneous closure of the left atrial appendage versus warfarin therapy for prevention of stroke in patients with atrial fibrillation: a randomised non-inferiority trial. Lancet. 2009 Aug 15;374(9689):534-42. doi: 10.1016/S0140-6736(09)61343-X. PMID 19683639
- [Background] Reddy VY, Doshi SK, Sievert H, Buchbinder M, Neuzil P, Huber K, Halperin JL, Holmes D; PROTECT AF Investigators. Percutaneous left atrial appendage closure for stroke prophylaxis in patients with atrial fibrillation: 2.3-Year Follow-up of the PROTECT AF (Watchman Left Atrial Appendage System for Embolic Protection in Patients with Atrial Fibrillation) Trial. Circulation. 2013 Feb 12;127(6):720-9. doi: 10.1161/CIRCULATIONAHA.112.114389. Epub 2013 Jan 16. PMID 23325525
- [Background] Kleinecke C, Gomez Monterrosas O, Scalone G, Lam YY, Shin ES, Bellmann B, Brachmann J, Park JW. First-in-human experience of left atrial appendage occlusion with the steerable FuStar sheath. J Interv Cardiol. 2018 Aug;31(4):532-537. doi: 10.1111/joic.12509. Epub 2018 Mar 26. PMID 29582475
- [Background] Huang H, Liu Y, Xu Y, Wang Z, Li Y, Cao K, Zhang S, Yang Y, Yang X, Huang D, Yu B, Su X, Wu L, Huang C. Percutaneous Left Atrial Appendage Closure With the LAmbre Device for Stroke Prevention in Atrial Fibrillation: A Prospective, Multicenter Clinical Study. JACC Cardiovasc Interv. 2017 Nov 13;10(21):2188-2194. doi: 10.1016/j.jcin.2017.06.072. PMID 29122133
- [Background] Park JW, Sievert H, Kleinecke C, Vaskelyte L, Schnupp S, Sievert K, Lam YY, Stahli BE, Zhang D, Li A, Brachmann J. Left atrial appendage occlusion with lambre in atrial fibrillation: Initial European experience. Int J Cardiol. 2018 Aug 15;265:97-102. doi: 10.1016/j.ijcard.2018.02.120. PMID 29885707
- [Background] Lansky AJ, Messe SR, Brickman AM, Dwyer M, van der Worp HB, Lazar RM, Pietras CG, Abrams KJ, McFadden E, Petersen NH, Browndyke J, Prendergast B, Ng VG, Cutlip DE, Kapadia S, Krucoff MW, Linke A, Moy CS, Schofer J, van Es GA, Virmani R, Popma J, Parides MK, Kodali S, Bilello M, Zivadinov R, Akar J, Furie KL, Gress D, Voros S, Moses J, Greer D, Forrest JK, Holmes D, Kappetein AP, Mack M, Baumbach A. Proposed Standardized Neurological Endpoints for Cardiovascular Clinical Trials: An Academic Research Consortium Initiative. J Am Coll Cardiol. 2017 Feb 14;69(6):679-691. doi: 10.1016/j.jacc.2016.11.045. PMID 28183511
- [Background] Mehran R, Rao SV, Bhatt DL, Gibson CM, Caixeta A, Eikelboom J, Kaul S, Wiviott SD, Menon V, Nikolsky E, Serebruany V, Valgimigli M, Vranckx P, Taggart D, Sabik JF, Cutlip DE, Krucoff MW, Ohman EM, Steg PG, White H. Standardized bleeding definitions for cardiovascular clinical trials: a consensus report from the Bleeding Academic Research Consortium. Circulation. 2011 Jun 14;123(23):2736-47. doi: 10.1161/CIRCULATIONAHA.110.009449. No abstract available. PMID 21670242
- [Background] VARC-3 WRITING COMMITTEE; Genereux P, Piazza N, Alu MC, Nazif T, Hahn RT, Pibarot P, Bax JJ, Leipsic JA, Blanke P, Blackstone EH, Finn MT, Kapadia S, Linke A, Mack MJ, Makkar R, Mehran R, Popma JJ, Reardon M, Rodes-Cabau J, Van Mieghem NM, Webb JG, Cohen DJ, Leon MB. Valve Academic Research Consortium 3: updated endpoint definitions for aortic valve clinical research. Eur Heart J. 2021 May 14;42(19):1825-1857. doi: 10.1093/eurheartj/ehaa799. PMID 33871579
- [Background] Robins JM, Finkelstein DM. Correcting for noncompliance and dependent censoring in an AIDS Clinical Trial with inverse probability of censoring weighted (IPCW) log-rank tests. Biometrics. 2000 Sep;56(3):779-88. doi: 10.1111/j.0006-341x.2000.00779.x. PMID 10985216
- [Background] Osmancik P, Herman D, Neuzil P, Hala P, Taborsky M, Kala P, Poloczek M, Stasek J, Haman L, Branny M, Chovancik J, Cervinka P, Holy J, Kovarnik T, Zemanek D, Havranek S, Vancura V, Opatrny J, Peichl P, Tousek P, Lekesova V, Jarkovsky J, Novackova M, Benesova K, Widimsky P, Reddy VY; PRAGUE-17 Trial Investigators. Left Atrial Appendage Closure Versus Direct Oral Anticoagulants in High-Risk Patients With Atrial Fibrillation. J Am Coll Cardiol. 2020 Jun 30;75(25):3122-3135. doi: 10.1016/j.jacc.2020.04.067. PMID 32586585
- [Background] Korsholm K, Damgaard D, Valentin JB, Packer EJS, Odenstedt J, Sinisalo J, Putaala J, Naess H, Al-Jazi MA, Karlsson JE, Pontoppidan J, Modrau B, Hjort J, Matzen KL, Johnsen SP, Nielsen-Kudsk JE. Left atrial appendage occlusion vs novel oral anticoagulation for stroke prevention in atrial fibrillation: rationale and design of the multicenter randomized occlusion-AF trial. Am Heart J. 2022 Jan;243:28-38. doi: 10.1016/j.ahj.2021.08.020. Epub 2021 Sep 17. PMID 34537184
- [Background] Sahay S, Nombela-Franco L, Rodes-Cabau J, Jimenez-Quevedo P, Salinas P, Biagioni C, Nunez-Gil I, Gonzalo N, de Agustin JA, Del Trigo M, Perez de Isla L, Fernandez-Ortiz A, Escaned J, Macaya C. Efficacy and safety of left atrial appendage closure versus medical treatment in atrial fibrillation: a network meta-analysis from randomised trials. Heart. 2017 Jan 15;103(2):139-147. doi: 10.1136/heartjnl-2016-309782. Epub 2016 Sep 1. PMID 27587437
- [Background] Cutlip DE, Windecker S, Mehran R, Boam A, Cohen DJ, van Es GA, Steg PG, Morel MA, Mauri L, Vranckx P, McFadden E, Lansky A, Hamon M, Krucoff MW, Serruys PW; Academic Research Consortium. Clinical end points in coronary stent trials: a case for standardized definitions. Circulation. 2007 May 1;115(17):2344-51. doi: 10.1161/CIRCULATIONAHA.106.685313. PMID 17470709
- [Background] Thygesen K, Alpert JS, Jaffe AS, Simoons ML, Chaitman BR, White HD; Writing Group on the Joint ESC/ACCF/AHA/WHF Task Force for the Universal Definition of Myocardial Infarction; Thygesen K, Alpert JS, White HD, Jaffe AS, Katus HA, Apple FS, Lindahl B, Morrow DA, Chaitman BA, Clemmensen PM, Johanson P, Hod H, Underwood R, Bax JJ, Bonow RO, Pinto F, Gibbons RJ, Fox KA, Atar D, Newby LK, Galvani M, Hamm CW, Uretsky BF, Steg PG, Wijns W, Bassand JP, Menasche P, Ravkilde J, Ohman EM, Antman EM, Wallentin LC, Armstrong PW, Simoons ML, Januzzi JL, Nieminen MS, Gheorghiade M, Filippatos G, Luepker RV, Fortmann SP, Rosamond WD, Levy D, Wood D, Smith SC, Hu D, Lopez-Sendon JL, Robertson RM, Weaver D, Tendera M, Bove AA, Parkhomenko AN, Vasilieva EJ, Mendis S; ESC Committee for Practice Guidelines (CPG). Third universal definition of myocardial infarction. Eur Heart J. 2012 Oct;33(20):2551-67. doi: 10.1093/eurheartj/ehs184. Epub 2012 Aug 24. No abstract available. PMID 22922414
- [Background] Korsholm K, Berti S, Iriart X, Saw J, Wang DD, Cochet H, Chow D, Clemente A, De Backer O, Moller Jensen J, Nielsen-Kudsk JE. Expert Recommendations on Cardiac Computed Tomography for Planning Transcatheter Left Atrial Appendage Occlusion. JACC Cardiovasc Interv. 2020 Feb 10;13(3):277-292. doi: 10.1016/j.jcin.2019.08.054. Epub 2019 Oct 30. PMID 31678086